CLINICAL TRIAL: NCT04015687
Title: A Phase 1, Open-label Study to Evaluate the Effect of AG-881 on the Pharmacokinetics of a Single Dose of Lamotrigine in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of AG-881 on the Pharmacokinetics of a Single Dose of Lamotrigine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AG881-C-006
Record Dates: First submitted 2019-07-03; First posted 2019-07-11 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Healthy Participants
Keywords: Pharmacokinetic study
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AG-881 (Group 1) (Experimental): On Day 1 of Period 1, Group 1 participants will receive a single 50-milligram (mg) oral dose of lamotrigine at Hour 0. In Period 2, they will receive 50-mg oral doses of AG-881 once daily (QD) for 15 consecutive days (Days 1 to 15), with a single 50-mg oral dose of lamotrigine coadministered at Hour 0 on Day 14.
  Interventions: Drug: AG-881; Drug: Lamotrigine
- AG-881 (Group 2) (Experimental): Following a safety and tolerability review of the data from at least 7 days of AG-881 dosing of Group 1 participants in Period 2, Group 2 participants will receive a single 50-mg oral dose of lamotrigine at Hour 0 in Period 1, and 50-mg oral doses of AG-881 QD for 15 consecutive days (Days 1 to 15), with a single 50-mg oral dose of lamotrigine coadministered at Hour 0 on Day 14 in Period 2.
  Interventions: Drug: AG-881; Drug: Lamotrigine
- AG-881 (Group 3) (Experimental): Following a safety and tolerability review of the data from Group 1 participants, and from at least 7 days of AG-881 dosing of Group 2 participants in Period 2, Group 3 participants will receive a single 50-mg oral dose of lamotrigine at Hour 0 in Period 1; and 50-mg oral doses of AG-881 QD for 15 consecutive days (Days 1 to 15) with a single 50-mg oral dose of lamotrigine coadministered at Hour 0 on Day 14 in Period 2.
  Interventions: Drug: AG-881; Drug: Lamotrigine

INTERVENTIONS:
Drug: AG-881 — Supplied as uncoated tablets.
Drug: Lamotrigine — Supplied as tablets of LAMICTAL® or generic equivalent.
  Other Names: LAMICTAL®

SUMMARY:
The main purpose of this study is to examine the effect of multiple doses of AG-881 on the pharmacokinetics (PK) of a single dose of lamotrigine in healthy adults.

ELIGIBILITY:
Inclusion criteria

* Healthy, adult, male or female participants, 18-55 years of age, inclusive, at screening;
* Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study, based on participant self-reporting;
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per square meter (kg/m^2) at screening;
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECG), as deemed by the principal investigator or designee;
* Liver function tests (serum alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase [ALP], and bilirubin [total and direct]) must be ≤ the upper limit of normal;
* Female participants must be of non-childbearing potential defined as a female who has undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

  * hysteroscopic sterilization;
  * bilateral tubal ligation or bilateral salpingectomy;
  * hysterectomy;
  * bilateral oophorectomy;
  * or is postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status;
* A non-vasectomized, male participant must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after the last dosing. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to the first dosing of study drug. A male who has been vasectomized less than 4 months prior to study first dosing must follow the same restrictions as a non-vasectomized male);
* If a male participant, must agree not to donate sperm from the first dosing until 90 days after the last dosing;
* Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion criteria:

* Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study;
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the principal investigator or designee;
* History of any illness that, in the opinion of the principal investigator or designee, might confound the results of the study or pose an additional risk to the participant (e.g., history or presence of rashes) by their participation in the study;
* History or presence of ventricular dysfunction or risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, cardiomyopathy, family history of Long QT Syndrome), in the opinion of the principal investigator or designee;
* History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing;
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds;
* Known medical history of progressive multifocal leukoencephalopathy;
* Presence of an active skin rash;
* Any positive responses on the Columbia-suicide severity rating scale (C-SSRS);
* Female participants of childbearing potential;
* Female participants with a positive pregnancy test or who are lactating;
* Positive urine drug or alcohol results at screening or first check-in;
* Positive results at screening for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies;
* Corrected QT interval by Fridericia (QTcF) is >450 milliseconds (msec), or Q wave, R wave, and S wave complex (QRS) interval >110 msec, or P wave to the start of the QRS complex (PR interval) >220 msec or participants who have ECG findings deemed abnormal with clinical significance by the principal investigator or designee at screening;
* Estimated creatinine clearance <90 millimeters per minute (mL/min) at screening;
* Unable to refrain from or anticipate the use of:

  * Any drug, including prescription and non-prescription medications, herbal remedies, and vitamin supplements, beginning 14 days prior to the first dosing and throughout the study. After first dosing, ibuprofen (1.2 grams [g] per 24 hours) may be administered at the discretion of principal investigator or designee;
  * Any drugs known to be strong inducers of cytochrome P450 (CYP) 3A enzymes or uridine 5´-diphospho-glucuronyl transferases (UGTs), including St. John's Wort, for 28 days prior to the first dosing and throughout the study. Appropriate sources (e.g., Flockhart Table™) will be consulted to confirm lack of pharmacokinetic/pharmacodynamic interaction with study drug;
* Refuses to abstain from grapefruit-containing foods or beverages or Seville orange containing foods or beverages from 14 days prior to the first dosing and throughout the study;
* Has been on a diet incompatible with the on-study diet, in the opinion of the principal investigator or designee, within the 30 days prior to the first dosing and throughout the study;
* Donation of blood or significant blood loss within 56 days prior to the first dose;
* Plasma donation within 7 days prior to the first dose;
* Participation in another clinical study within 30 days prior to the first dose. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Area under the Concentration-time Curve from Time 0 to Infinity (AUC0-inf) for Lamotrigine Administered with Interacting Drug AG-881 | At multiple time points daily from Day 14 to Day 21 (or early discontinuation) in Period 2 (21-day period)
Area under the Concentration-time Curve from Time 0 to Infinity (AUC0-inf) for Lamotrigine Administered without Interacting Drug AG-881 | At multiple time points daily from Day 1 to Day 8 in Period 1 (8-day period)
Maximum Observed Plasma Concentration (Cmax) for Lamotrigine Administered with Interacting Drug AG-881 | At multiple time points daily from Day 14 to Day 21 (or early discontinuation) in Period 2 (21-day period)
Maximum Observed Plasma Concentration (Cmax) for Lamotrigine Administered without Interacting Drug AG-881 | At multiple time points daily from Day 1 to Day 8 in Period 1 (8-day period)
Area under the Concentration-time Curve, from Time 0 to the Last Observed Non-zero Concentration (t) (AUC0-t) for Lamotrigine Administered with Interacting Drug AG-881 | At multiple time points daily from Day 14 to Day 21 (or early discontinuation) in Period 2 (21-day period)
Area under the Concentration-time Curve, from Time 0 to the Last Observed Non-zero Concentration (t) (AUC0-t) for Lamotrigine Administered without Interacting Drug AG-881 | At multiple time points daily from Day 1 to Day 8 in Period 1 (8-day period)
Percent of AUC0-inf Extrapolated (AUC%extrap) for Lamotrigine Administered with Interacting Drug AG-881 | At multiple time points daily from Day 14 to Day 21 (or early discontinuation) in Period 2 (21-day period)
Percent of AUC0-inf Extrapolated (AUC%extrap) for Lamotrigine Administered without Interacting Drug AG-881 | At multiple time points daily from Day 1 to Day 8 in Period 1 (8-day period)
Time to Maximum Observed Plasma Concentration (Tmax) for Lamotrigine Administered with Interacting Drug AG-881 | At multiple time points daily from Day 14 to Day 21 (or early discontinuation) in Period 2 (21-day period)
Time to Maximum Observed Plasma Concentration (Tmax) for Lamotrigine Administered without Interacting Drug AG-881 | At multiple time points daily from Day 1 to Day 8 in Period 1 (8-day period)
Apparent Terminal Elimination Rate Constant (Kel) for Lamotrigine Administered with Interacting Drug AG-881 | At multiple time points daily from Day 14 to Day 21 (or early discontinuation) in Period 2 (21-day period)
Apparent Terminal Elimination Rate Constant (Kel) for Lamotrigine Administered without Interacting Drug AG-881 | At multiple time points daily from Day 1 to Day 8 in Period 1 (8-day period)
Apparent Terminal Elimination Half-life (t½) for Lamotrigine Administered with Interacting Drug AG-881 | At multiple time points daily from Day 14 to Day 21 (or early discontinuation) in Period 2 (21-day period)
Apparent Terminal Elimination Half-life (t½) for Lamotrigine Administered without Interacting Drug AG-881 | At multiple time points daily from Day 1 to Day 8 in Period 1 (8-day period)
Apparent Total Plasma Clearance after Oral (Extravascular) Administration (CL/F) for Lamotrigine Administered with Interacting Drug AG-881 | At multiple time points daily from Day 14 to Day 21 (or early discontinuation) in Period 2 (21-day period)
Apparent Total Plasma Clearance after Oral (Extravascular) Administration (CL/F) for Lamotrigine Administered without Interacting Drug AG-881 | At multiple time points daily from Day 1 to Day 8 in Period 1 (8-day period)
Apparent Volume of Distribution during the Terminal Elimination Phase after Oral (Extravascular) Administration (Vz/F) for Lamotrigine Administered with Interacting Drug AG-881 | At multiple time points daily from Day 14 to Day 21 (or early discontinuation) in Period 2 (21-day period)
Apparent Volume of Distribution during the Terminal Elimination Phase after Oral (Extravascular) Administration (Vz/F) for Lamotrigine Administered without Interacting Drug AG-881 | At multiple time points daily from Day 1 to Day 8 in Period 1 (8-day period)

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to approximately 4 weeks
  An AE is any untoward medical occurrence associated with the use of a drug, whether or not considered drug-related.
Columbia-suicide Severity Rating Scale (C-SSRS) | Up to approximately 4 weeks
  The C-SSRS is a questionnaire scale to detect emergent suicide symptoms (suicidal ideation or actual suicidal behavior). Questions are either answered yes/no or are on a scale of 1 (low severity) to 5 (high severity).
Percentage of Participants with Abnormalities in 12-lead Electrocardiograms (ECGs) | Up to approximately 4 weeks
Percentage of Participants with Abnormalities in Vital Sign Measurements | Up to approximately 4 weeks
  Vital signs will include body temperature, respiratory rate, blood pressure, and heart rate.
Percentage of Participants with Abnormalities in Clinical Laboratory Tests | Up to approximately 4 weeks
  Clinical laboratory assessments will include hematology, serum chemistry, coagulation, and urinalysis.
Percentage of Participants with Abnormalities in Physical Examinations | Up to approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Agios Pharmaceuticals, Inc.
Locations (1):
- Celerion, Inc, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No